CLINICAL TRIAL: NCT07135895
Title: The Artix All-in-one Solution for Complete thrombEctomy With eNDovascular Approach
Brief Title: The ArtixASCEND Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-001
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Lower Limb Arterial Occlusion
Keywords: Acute Limb Ischemia; Lower limb arterial occlusion; Artix Thrombectomy System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Artix Thrombectomy System (Experimental): Non-surgical removal of lower extremity arterial emboli and thrombi using the Artix Thrombectomy System.
  Interventions: Device: Artix Thrombectomy System

INTERVENTIONS:
Device: Artix Thrombectomy System — Treatment of lower extremity arterial occlusions using the Artix Thrombectomy System.

SUMMARY:
This study is a post-market, prospective, multicenter, single-arm study to evaluate the safety and effectiveness of the Artix Thrombectomy System in patients with acute lower extremity arterial occlusions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute symptom duration ≤ 14 days
* Lower limb arterial occlusion below inguinal ligament
* Target lesion in native vessel
* Target vessel size between 3 mm and 8 mm by visual estimation
* Rutherford category I, IIa, or IIb
* Informed consent is obtained from either patient or legally authorized representative (LAR) per Institutional Review Board/Ethics Committee requirements

Exclusion Criteria:

* Life expectancy < 6 months
* Prior major amputation in the target limb
* Prior minor amputation in the target limb that is not completely healed or cannot bear weight
* Non-thrombotic occlusion secondary to dissection, vasculitis, or target vessel trauma
* Treatment of the index event in the target vessel with any other endovascular thrombectomy/aspiration or open surgical method prior to Artix procedure
* Part of a vulnerable population (e.g., currently pregnant, breastfeeding or incarcerated) per local definitions
* Known sensitivity to radiographic contrast agents that, in the Investigator's opinion, cannot be adequately pre-treated
* Unable to tolerate antiplatelet therapy
* Inability to anticoagulate the patient with heparin, enoxaparin or other parenteral antithrombin, or known to have uncorrected bleeding disorders (e.g., gastro-intestinal ulcer, menorrhagia, liver failure, heparin-induced thrombocytopenia (HIT))
* Any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject (e.g., contraindication to use of Artix per local approved labeling, compromise the well-being or that could prevent, limit, or confound the protocol-specified assessments)
* Current participation in another drug or device study that, in the investigator's opinion, would interfere with participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | Immediately Following Index Procedure
  Revascularization rate post-index procedure of target treatment area determined by an independent core lab.
Primary Safety Endpoint | 48 Hours
  Periprocedural (within 48 hours) Artix Thrombectomy System-related major bleeding rate adjudicated as causal to the study device as determined by an independent Medical Monitor.

SECONDARY OUTCOMES:
Distal embolization SAEs | Intra-procedure
All-cause mortality | 1-month follow-up visit
Limb salvage | 1-month follow-up visit
  Freedom from major amputation of the index limb
Amputation-free survival | 1-month follow-up visit
  Freedom from major amputation and all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh Willson, Study Director — Inari Medical

IPD SHARING:
Plan to Share IPD: No